CLINICAL TRIAL: NCT03541954
Title: Neurophysiological Validation of the Clinical Criteria of Sensitization in Chronic Pelvic and Perineal Pain Population : a Prospective Controlled Interventional Study
Brief Title: Neurophysiological Validation of the Clinical Criteria of Sensitization in Chronic Pelvic and Perineal Pain Population
Acronym: DOPEC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of inclusions
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: RC17_0427
Record Dates: First submitted 2018-05-17; First posted 2018-05-31 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Chronic Pelvic Pain; Chronic Perineal Pain
Keywords: sensitization; pain thresholds

STUDY DESIGN:
Intervention Model Description: 2 types of patients will be included:
  * 30 patients with chronic pelvic or perineal pain with sensitization (Convergences PP criteria > 5)
  * 30 patients with chronic pelvic or perineal pain without sensitization (Convergences PP criteria < 5)
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with pelvic or perineal pain with sensitization (Other): Patients with chronic pelvic or perineal pain with sensitization (Convergences PP criteria > 5)
  Interventions: Other: Sensory testing of lower urinary tract.; Other: Sensory testing of lower rectal tract; Other: Sensory testing of vulva muscles; Other: Sensory testing of pelvic muscles
- Patient with pelvic or perineal pain without sensitization (Other): Patients with chronic pelvic or perineal pain without sensitization (Convergences PP criteria < 5)
  Interventions: Other: Sensory testing of lower urinary tract.; Other: Sensory testing of lower rectal tract; Other: Sensory testing of vulva muscles; Other: Sensory testing of pelvic muscles

INTERVENTIONS:
Other: Sensory testing of lower urinary tract. — Non invasive lower urinary tract sensitivity testing: provoked diuresis with sonographic estimates of sensory thresholds.
Other: Sensory testing of lower rectal tract — Lower digestive tract sensitivity testing: rectal electronic barostat with ascending pressure (phasic distension).
Other: Sensory testing of vulva muscles — Vulvar sensitivity testing: pressure pain threshold evaluated using vulvagesiometer.
Other: Sensory testing of pelvic muscles — Myofascial sensitivity testing: piriformis, levator ani and obturator internus muscles pressure pain threshold evaluated using intra-vaginal algometer.

SUMMARY:
The purpose of this study is to assess and validate the clinical criteria of sensitization ("Convergences PP criteria") selected by the expert consensus with neurophysiological sensory testing.

DETAILED DESCRIPTION:
Some patient with chronic pelvic or perineal pain, present complex manifestations, comprising pain and dysfunction which does not involved a single organ. The gap between clinical symptoms and pathological signs is a constant feature of these pain syndromes. A possible explanation for these pain syndromes is central sensitization. This sensitization is defined by decrease nociceptive thresholds, a more intense and more prolonged response to nociceptive stimulus, and spatial extension of the painful area. It has been defined by international expert consensus in 2016 a clinical evaluation tool with 10 criteria for sensitization diagnosis: Convergences PP criteria. The aim of this study is to objectivize lower threshold, spatial and temporal diffusion of pain in women with chronic pelvic or perineal pain with sensitization (Convergences PP criteria > 5) compared to women without sensitization (Convergences PP criteria < 5). A sensory testing of lower urinary tract, lower rectal tract, vulva and pelvic muscles will be achieved.

ELIGIBILITY:
Inclusion Criteria:

* Women > 25 years,
* Pelvic or perineal pain since > 3 months,
* No injury in pelvic imagery or clinical examination that may explain all the pain complaint,
* Patient who can understand the protocol,
* Patient who agreed and signed the informed consent for participation.

Exclusion Criteria:

* Poor understanding of French language,
* Pregnancy or lactation,
* Severe depression (Beck Depression Inventory-Short form > 16),
* Initial pain estimation at 10 on numeric analog scale,
* Inadequately cooperating,
* Isolated dysmenorrhea,
* Deep endometriosis with rectal or bladder lesion,
* Genital or bladder infection,
* Urogenital tumor history,
* Anorectal surgery history a type of digestive resection,
* Anal stenosis,
* Advanced vaginal prolapse (stage 2 on POP-Q scale),
* Post-traumatic stress disorder history,
* Deprived of liberty (trusteeship, guardianship).

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Comparison of pelvic pain threshold | 1 month after inclusion in the study
  Comparison of pelvic pain threshold obtained by 4 neurophysiological testing, between women with chronic pelvic or perineal pain with sensitization (Convergences PP criteria > 5) and without sensitization (Convergences PP criteria < 5).

SECONDARY OUTCOMES:
Identification of temporal distribution of pain | 1 month after inclusion in the study
  Identification of temporal distribution of pain in women with chronic pelvic or perineal pain with sensitization (Convergences PP criteria > 5) compared to women without sensitization (Convergences PP criteria < 5).
Identification of lower pain perception thresholds | 1 month after inclusion in the study
  Identification of lower pain perception thresholds in women with chronic pelvic or perineal pain with sensitization (Convergences PP criteria > 5) compared to women without sensitization (Convergences PP criteria < 5) for each of the 4 neurophysiological testing.
Comparison of state anxiety | 1 month after inclusion in the study
  Comparison of state anxiety between women with chronic pelvic or perineal pain with sensitization (Convergences PP criteria > 5) and without sensitization (Convergences PP criteria < 5).
Comparison of depression | 1 month after inclusion in the study
  Comparison of depression between women with chronic pelvic or perineal pain with sensitization (Convergences PP criteria > 5) and without sensitization (Convergences PP criteria < 5).
Comparison of catastrophizing | 1 month after inclusion in the study
  Comparison of catastrophizing between women with chronic pelvic or perineal pain with sensitization (Convergences PP criteria > 5) and without sensitization (Convergences PP criteria < 5).
Comparison of quality of life | 1 month after inclusion in the study
  Comparison of quality of life between women with chronic pelvic or perineal pain with sensitization (Convergences PP criteria > 5) and without sensitization (Convergences PP criteria < 5).

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Nantes university Hospital, Nantes
  - Groupe Confluent, Nantes

REFERENCES:
- [Derived] Cardaillac C, Levesque A, Riant T, Mortier A, Neunlist M, Perrouin-Verbe MA, Volteau C, Thubert T, Brochard C, Ploteau S. Evaluation of a scoring system for the detection of central sensitization among women with chronic pelvic pain. Am J Obstet Gynecol. 2023 Nov;229(5):530.e1-530.e17. doi: 10.1016/j.ajog.2023.07.044. Epub 2023 Jul 27. PMID 37516398